CLINICAL TRIAL: NCT04932018
Title: Exploring the Feasibility of a Start-up Incubator to Decrease Occupational Stress and Depression in Beginning Kentucky Farmers
Brief Title: Exploring an Incubator to Decrease Stress in Farmers Occupational Stress and Depression in Beginning Kentucky Farmers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Martha Biddle (Other)
Collaborators: National Institute for Occupational Safety and Health (NIOSH/CDC) (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Martha Biddle, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 61320
Record Dates: First submitted 2021-06-10; First posted 2021-06-18 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Occupational Stress; Depression
MeSH Terms: conditions — Occupational Stress; Depression

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (Experimental): The intervention group will participate in a round table educational session with a study facilitator/mentor farmer and occupational health nurse plus receive an invitation to participate in an interactive virtual community providing ongoing resources and support from community farmers and agriculture experts.
  Interventions: Behavioral: Virtual Community of Support; Behavioral: Mentorship Incubator
- Attention Control (Sham Comparator): The second group (attention control) will receive an invitation to participate in the virtual community without mentor interaction.
  Interventions: Behavioral: Virtual Community of Support

INTERVENTIONS:
Behavioral: Virtual Community of Support — The 6-month virtual community will consist of self-directed learning modules that will vary in content from worker and family relationships, collaboration and skill acquisition to self-care habits; problem-solving; monthly sessions will include a positive psychology exercise.
Behavioral: Mentorship Incubator — The 6-month incubator intervention will consist of monthly interactive time with an assigned study facilitator/farmer mentor.
  Arms: Interventional

SUMMARY:
The purpose of this 6- month study is to determine the feasibility of a start-up incubator intervention designed to decrease occupational stress and depression for beginning Kentucky farmers. The objectives are to: #1) test the feasibility of a mentorship and start-up incubator intervention on depression in beginning Kentucky farmers using questionnaires administered prestudy, mid-study, and post-study; #2) explore associations between mentorship, occupational stress and depression in beginning Kentucky farmers using specific survey questionnaires to guide future research. This study's results will provide valuable data to agriculture and occupational health researchers. The data will illustrate the impact of mentorship and community support on improving depression and occupational stress of beginning Kentucky farmers.

DETAILED DESCRIPTION:
A suicide rate in farmers which is higher than the general population (rate 17.3/100,000) should remind occupational health professionals that the important work of agriculture is creating an emotional burden resulting in preventable death. Given the high incidence of suicide in the farming population, it is imperative that we explore the agrarian culture to guide the development of interventions to reduce occupational stress and depression in beginning Kentucky farmers. The isolating nature of rural farming, a leading risk factor for depression, creates an urgency to develop interventions to protect our Kentucky farmers from occupational stress and depression, which are leading risk factors for suicide. Interventions developed to reduce occupational stress and depression are an essential strategy to improve mental health before the devastating outcome of suicide. To address a gap in the management of occupational stress and depression in beginning farmers in Kentucky, novel interventions must address the unique agrarian culture, rural isolation, peer influence and social stigma of depression. Interventions must be available at little to no expense and without extensive time commitment; must be accessible in rural areas and provide mentorship and community support. The concept of a start-up incubator for beginning farmers is one type of intervention that combines the accessibility of a virtual program with mentorship by farming experts, peer and community support, with a mental health curriculum provided by occupational health nurses is our proposed intervention to address occupational stress and depression in the beginning Kentucky farmer. The curriculums of several existing programs related to occupational stress and depression guide the development of this incubator intervention. Incubator curriculums are designed to address failures and mitigate conditions to support future success. Rural Resilience, Farm Aid, and Farm Stress are training programs that address stress, depression, and suicide in farmers, these programs use components of an incubator model to fit the constructs of agrarian business and culture. The start-up incubator model in this proposal utilizes mentorship and community support to form a strategic alliance between mentors and beginner farmers.

Mentorship and community support are social capital that can be utilized through networking opportunities which may eliminate the structural barriers identified by beginning farmers. The impact of mentorship and community support in the context of healthcare, business, and farming has consistently been supported in research. Uncomfortable topics of occupational stressors and depression have only recently been included in initiatives to help farmers, however available mentorship programs in Kentucky are currently focused on farm management knowledge deficits. Results from this proposed study have the potential to guide future research related to the effectiveness for occupational stress, depression and suicide reduction in beginning Kentucky farmers. This proposal will address a major mental health objective of Healthy People 2020: Reducing the rising national suicide rate, specifically by addressing the vulnerable population of farmworkers considered to be at high risk (https://www.healthypeople.gov/node/4804/data_details). The The purpose of this study is to determine the feasibility of a start-up incubator intervention designed to decrease occupational stress and depression for beginning Kentucky farmers. The central hypothesis is: A start-up incubator intervention will be feasible and acceptable to the beginning farmer population. Specific Aim #1: To test the feasibility of a start-up incubator intervention on occupational stress and depression in beginning Kentucky farmers. Hypothesis #1: Compared to an attention control group, individuals assigned to the incubator intervention (6 month curriculum) group will have a lower incidence of occupational stress and depression at three and six months from baseline.

Specific Aim #2: To explore associations between mentorship, occupational stress and depression in beginning Kentucky farmers to guide future research. Hypothesis #2: Associations exist between mentorship, occupational stress and depression that will guide future research focused on prioritizing efforts to advance farmer health and well-being.

Study Design. The design is that of a two-group intervention study. Subjects (N=48) will be assigned to 1 of 2 groups (intervention group or attention control group based on county of residence; randomization will occur at the county level). Subjects will be recruited from eight central Kentucky counties: Washington, Anderson, Franklin, Henry, Scott, Harrison, Woodford and Owen. The intervention group will participate in a round table educational session with a study facilitator/mentor farmer and occupational health nurse plus receive an invitation to participate in an interactive virtual community providing ongoing resources and support from community farmers and agriculture experts. The second group (attention control) will receive an invitation to participate in the virtual community without mentor interaction. Data collection for both groups will occur at baseline, 3 months, and 6-months.

Sample and Setting. Subjects will be referred by county extension agents located in Washington, Anderson, Franklin, Henry, Scott, Harrison, Woodford and Owen counties in Kentucky that have contact with "beginning farmers", as defined by the United States Department of Agriculture (USDA). Subjects will be contacted via email or personal contact by County Extension agents, or via CCTS recruitment services, potential interested parties will be given the PI's email, name and phone to contact for pre-screening of eligibility into the study. A total of 48 subjects meeting inclusion criteria will be assigned to one of two groups. Based on USDA estimates of beginning farmer characteristics, the planned enrollment in this study is 60% men, 95% Caucasian, and 5% Black or African American (demographic survey will include a question regarding Hispanic ethnicity).

ELIGIBILITY:
Inclusion Criteria:

* classified as a beginning farmer by the USDA criteria
* has the ability to read and speak English;
* access to wi-fi or smartphone technology.
* primary residence or farm in Washington, Anderson, Franklin, Henry, Scott, Harrison, Woodford or Owen County, Kentucky

Exclusion Criteria:

- less than 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Occupational Stress | Change from baseline occupational stress at 6 months
  Psychological stress as result of farming measured with the Farm Stressors Inventory, a 37 item self-report survey measuring potentially prevalent farm stressors. Items from the following categories of stressors are addressed in the assessment tool: personal finances, weather, regulatory climate, workload and other job demands, physical environment, control and ambiguity, interpersonal issues, and job and retirement security. The tool is comprised of a 1-5 likert scale of 37 items, higher scores indicating higher occupational stress related to farming.
Depressive symptoms | Change from baseline depressive symptoms at 6 months
  Depressive symptoms as measured with the 10-item short Beck Depression Inventory to detect moderate and severe depressive episodes. High sensitivity and negative predictive value (NPV) were obtained with a cut-off score of 9/10 (sensitivity = 100%, specificity = 83.1%, NPV = 100%). High sensitivity and positive predictive value (PPV) were obtained with a cut-off score of 13/14 (sensitivity = 93.5%, specificity = 96%, PPV = 85.3%). The area under the ROC curve was 98.4% (95% Confidence Interval = 0.97-1.00). This tool includes 10 items, each including four alternative statements ranging in order of severity from zero to three. For the short form ,higher scores indicate higher depression.

SECONDARY OUTCOMES:
Self-Efficacy | Change from baseline self-efficacy at 6 months
  Self-efficacy will be measured with the John Henry Active Coping Scale, a 12 item self-report survey measuring coping strategies associated with sustained cognitive and emotional stressors. The scale includes twelve items answered on a Likert Scale with responses ranging from 1 "completely false" to 5 "completely true." Sample items include, "hard work has really helped me to get ahead"; "it's not always easy, but I manage to find a way to do the things I really need to get done"; and "once I make up my mind to do something, I stay with it until the job is completely done." The items were summed, with higher scores indicating a higher degree of high-effort coping
Adherence to Intervention | 6 months
  Intervention fidelity will be monitored by the PI, who will ensure all research assistants and study facilitators follow the study protocol. Study participants assigned to the intervention will have adherence monitored by participation in the virtual community and at the face to face meeting.

CONTACTS AND LOCATIONS:
Overall Officials: Martha Biddle, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Olson KR, Schellenberg RP. Farm stressors. Am J Community Psychol. 1986 Oct;14(5):555-69. doi: 10.1007/BF00935358. PMID 3799552
- [Background] Cuthbertson C, Brennan A, Shutske J, Zierl L, Bjornestad A, Macy K, Schallhorn P, Shelle G, Dellifield J, Leatherman J, Lin E, Skidmore M. Developing and Implementing Farm Stress Training to Address Agricultural Producer Mental Health. Health Promot Pract. 2022 Jan;23(1):8-10. doi: 10.1177/1524839920931849. Epub 2020 Jun 9. PMID 32517517
- [Background] Gerrard N. An application of a community psychology approach to dealing with farm stress. Can J Commun Ment Health. 2000 Fall;19(2):89-100. doi: 10.7870/cjcmh-2000-0017. PMID 11381740
- [Background] Hoyt DR, Conger RD, Valde JG, Weihs K. Psychological distress and help seeking in rural America. Am J Community Psychol. 1997 Aug;25(4):449-70. doi: 10.1023/a:1024655521619. PMID 9338954
- [Background] Peterson C, Stone DM, Marsh SM, Schumacher PK, Tiesman HM, McIntosh WL, Lokey CN, Trudeau AT, Bartholow B, Luo F. Suicide Rates by Major Occupational Group - 17 States, 2012 and 2015. MMWR Morb Mortal Wkly Rep. 2018 Nov 16;67(45):1253-1260. doi: 10.15585/mmwr.mm6745a1. PMID 30439869
- [Background] Cassitto MG, Gilioli R. [Emerging aspects of occupational stress]. Med Lav. 2003 Jan-Feb;94(1):108-13. Italian. PMID 12768962
- [Background] Oatley K, Bolton W. A social-cognitive theory of depression in reaction to life events. Psychol Rev. 1985 Jul;92(3):372-88. No abstract available. PMID 4023147
- [Background] Rudolphi JM, Berg RL, Parsaik A. Depression, Anxiety and Stress Among Young Farmers and Ranchers: A Pilot Study. Community Ment Health J. 2020 Jan;56(1):126-134. doi: 10.1007/s10597-019-00480-y. Epub 2019 Oct 3. PMID 31583619
- [Background] Frey LM, Hans JD, Cerel J. Perceptions of Suicide Stigma. Crisis. 2016 Mar;37(2):95-103. doi: 10.1027/0227-5910/a000358. Epub 2015 Dec 23. PMID 26695868
- [Background] Kris-Etherton PM, Petersen KS, Hibbeln JR, Hurley D, Kolick V, Peoples S, Rodriguez N, Woodward-Lopez G. Nutrition and behavioral health disorders: depression and anxiety. Nutr Rev. 2021 Feb 11;79(3):247-260. doi: 10.1093/nutrit/nuaa025. PMID 32447382
- [Background] Logstein B. Farm-Related Concerns and Mental Health Status Among Norwegian Farmers. J Agromedicine. 2016;21(4):316-26. doi: 10.1080/1059924X.2016.1211055. PMID 27420178
- [Background] Hammen C. Stress and depression. Annu Rev Clin Psychol. 2005;1:293-319. doi: 10.1146/annurev.clinpsy.1.102803.143938. PMID 17716090
- [Background] Truchot D, Andela M. Burnout and hopelessness among farmers: The Farmers Stressors Inventory. Soc Psychiatry Psychiatr Epidemiol. 2018 Aug;53(8):859-867. doi: 10.1007/s00127-018-1528-8. Epub 2018 May 3. PMID 29725701
- [Background] Fernander AF, Duran RE, Saab PG, Llabre MM, Schneiderman N. Assessing the reliability and validity of the John Henry Active Coping Scale in an urban sample of African Americans and white Americans. Ethn Health. 2003 May;8(2):147-61. doi: 10.1080/13557850303563. PMID 14671768

DOCUMENTS (1):
  • Informed Consent Form (2022-03-07): https://cdn.clinicaltrials.gov/large-docs/18/NCT04932018/ICF_000.pdf